CLINICAL TRIAL: NCT06699641
Title: Cmparison Between the Kampala Trauma Score and the Estimated Injury Severity Score in the Outcome of Polytrauma Patients in the Emergency Departments in Egypt.
Brief Title: The Kampala Trauma Score in the Outcome of Polytrauma Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdallah Sayed Sawy, Resident, Assiut University
Other Study IDs: The Kampala Trauma Score value
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Polytrauma Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn about the predictive value of the Kampala Trauma Score in Egypt.

The main question it aims to answer is:

How does the performance of the Kampala Trauma Score compare to the Estimated Injury Severity Score in predicting outcomes for multi-traumatic patients in Egypt? Participants are adult polytrauma patients admitted to the emergency department during the study period.

DETAILED DESCRIPTION:
Two prominent scoring systems used in trauma care are the Kampala Trauma Score (KTS) and the Estimated Injury Severity Score (EISS). The KTS was specifically designed for use in low-resource settings, offering a practical tool for predicting patient outcomes based on readily available clinical data. This score integrates parameters such as age, systolic blood pressure, and Glasgow Coma Scale (GCS) scores, making it suitable for environments where advanced diagnostic tools may be lacking. Previous research has demonstrated the KTS's utility in various resource-limited settings, highlighting its role in effectively stratifying trauma patients and guiding triage decisions.

In contrast, the Estimated Injury Severity Score (EISS) is an adaptation of the Injury Severity Score (ISS), which incorporates both clinical and radiographic data to assess trauma severity comprehensively. The EISS uses an estimated approach to account for the often incomplete or preliminary information available in some clinical settings, aiming to provide a robust prediction of patient outcomes. While it is a more comprehensive tool than the KTS, its reliance on advanced imaging and detailed clinical information may limit its applicability in settings with restricted resources.

This study aims to conduct a cross-sectional comparison of the KTS and EISS to evaluate their relative effectiveness in assessing trauma severity and predicting patient outcomes. The results will provide valuable insights into the optimal use of trauma scoring systems and potentially inform improvements in trauma care practices

ELIGIBILITY:
Inclusion Criteria:

* Adult polytrauma patients
* Both genders

Exclusion Criteria:

* Patients with incomplete data or those who decline participation.
* Patients with multiple comorbidities.
* Patients managed outside the hospital.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Polytrauma patients admitted to the emergency departments at Assiut University Hospital located in Assiut/Egypt and Suez Canal University Hospital located in Ismailia/Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Outcome of polytrauma patients as assessed by the Kampala Trauma Score | From admission to 24 hours post admission
  From 0 to 10 9-10 = mild 7-8 = moderate <6 = severe

IPD SHARING:
Plan to Share IPD: No